CLINICAL TRIAL: NCT02985879
Title: A Randomized, Double-Blind, Placebo-Controlled Multiple Dose Study to Assess Efficacy, Safety, Tolerability, and Pharmacokinetics of ABBV-8E12 in Progressive Supranuclear Palsy
Brief Title: A Study to Assess Efficacy, Safety, Tolerability, and Pharmacokinetics of ABBV-8E12 in Subjects With Progressive Supranuclear Palsy (PSP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was prematurely discontinued because the program for progressive supranuclear palsy was discontinued due to lack of efficacy of study drug.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-562; 2016-001635-12 (EudraCT Number)
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Progressive Supranuclear Palsy
Keywords: PSP; Steele-Richardson-Olszewski syndrome; Tauopathy
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Tauopathies | interventions — tilavonemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): 0.9% Sodium Chloride Injection/Solution for Infusion; intravenous infusions at Day 1, Day 15, and Day 29, then every 28 days for 52 weeks
  Interventions: Drug: Placebo
- ABBV-8E12 2000 mg (Experimental): Intravenous infusions at Day 1, Day 15, and Day 29, then every 28 days for 52 weeks; 300 mg/15 mL (participants in countries other than Japan or Spain); 1000 mg/10 mL (for participants in Japan or Spain)
  Interventions: Drug: ABBV-8E12
- ABBV-8E12 4000 mg (Experimental): Intravenous infusions at Day 1, Day 15, and Day 29, then every 28 days for 52 weeks; 300 mg/15 mL (participants in countries other than Japan or Spain); 1000 mg/10 mL (for participants in Japan or Spain)
  Interventions: Drug: ABBV-8E12

INTERVENTIONS:
Drug: Placebo — Participants with 44-49 kg body weight (BW) had an intravenous infusion rate of 3.5 mL/min or 210 mL/hr; those with 50-58 kg BW, 4.0 mL/min or 240 mL/hr; and those with a BW >59 kg, 4.7 mL/min or 282 mL/hr.
  Arms: Placebo
Drug: ABBV-8E12 — Participants with 44-49 kg body weight (BW) had an intravenous infusion rate of 3.5 mL/min or 210 mL/hr; those with 50-58 kg BW, 4.0 mL/min or 240 mL/hr; and those with a BW >59 kg, 4.7 mL/min or 282 mL/hr. For participants in Cohort 2, ABBV-8E12 doses may have been decreased after the evaluation by the Data Monitoring Committee of available safety, tolerability and pharmacokinetic data.
  Other Names: Tilavonemab
  Arms: ABBV-8E12 2000 mg; ABBV-8E12 4000 mg

SUMMARY:
The purpose of this study was to assess efficacy, safety, tolerability, and pharmacokinetics of ABBV-8E12 in participants with progressive supranuclear palsy (PSP).

DETAILED DESCRIPTION:
This was a Phase 2, randomized, double-blind, placebo-controlled, multiple dose, multicenter study consisting of a screening period of up to 8 weeks (56 days), a 52-week double-blind treatment period, and a post-treatment follow-up period of approximately 20 weeks following last study drug administration (for those participants who prematurely discontinued from treatment, declined to participate in or did not qualify for participation in a long term extension [LTE] study). At the end of the treatment period, extended treatment was available for eligible participants who completed the 52-week treatment period and entered the separate long-term extension study (NCT03391765; Study M15-563). There were 3 cohorts in the study (Cohort 1, Cohort J1, and Cohort 2). Cohort 1 had augmented safety and pharmacokinetic (PK) assessments in the first 30 participants enrolled into the global study from countries other than Japan. Cohort J1 had augmented safety and PK assessments in the first 9 participants enrolled into the study from Japan. Cohort 2 consisted of all other participants enrolled in the global study not participating in Cohort 1 or Cohort J1.

This study was prematurely discontinued because the program for progressive supranuclear palsy was discontinued due to lack of efficacy of study drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participant with age 40 years or greater at the time of signed consent
* Meets the criteria for possible or probable progressive supranuclear palsy (PSP; Steele-Richardson-Olszewski Syndrome)
* Presence of PSP symptoms for less than 5 years
* Participant is able to walk 5 steps with minimal assistance (stabilization of one arm or use of cane/walker)
* Participant has an identified, reliable, study partner (e.g., caregiver, family member, social worker, or friend)

Key Exclusion Criteria:

* Participants who weigh less than 44 kg (97 lbs) at screening
* Mini-Mental State Examination (MMSE) score less than 15 at screening
* Any contraindication or inability to tolerate brain magnetic resonance imaging (MRI)
* Participant resides at a skilled nursing or dementia care facility, or admission to such a facility is planned during the study period
* Evidence of any clinically significant neurological disorder other than PSP
* The participant has a history of or currently has schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) or International Classification of Diseases (ICD-10) criteria
* Participant has had a significant illness or infection requiring medical intervention in the past 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (66):
- United States (27):
  - University of Alabama at Birmingham - Main /ID# 144892, Birmingham, Alabama
  - Mayo Clinic - Scottsdale /ID# 144893, Scottsdale, Arizona
  - Cedars-Sinai Medical Center /ID# 149775, Beverly Hills, California
  - Ucsd /Id# 144905, La Jolla, California
  - Usc /Id# 149773, Los Angeles, California
  - University of California, Los Angeles /ID# 144896, Los Angeles, California
  - Univ California, San Francisco /ID# 144897, San Francisco, California
  - Rocky Mountain Movement Disorders Center /ID# 153397, Englewood, Colorado
  - University of Florida - Archer /ID# 144906, Gainesville, Florida
  - Mayo Clinic /ID# 144911, Jacksonville, Florida
  - University of South Florida /ID# 144912, Tampa, Florida
  - Georgia Regents University /ID# 144908, Augusta, Georgia
  - Rush University Medical Center /ID# 144894, Chicago, Illinois
  - University of Chicago /ID# 148672, Chicago, Illinois
  - Indiana University /ID# 149036, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center /ID# 144891, Lexington, Kentucky
  - Mayo Clinic - Rochester /ID# 144895, Rochester, Minnesota
  - St. Luke's Hosp. of Kansas Cit /ID# 168629, Kansas City, Missouri
  - Cleveland Clinic Lou Ruvo Cent /ID# 148919, Las Vegas, Nevada
  - Rutgers Robert Wood Johnson /ID# 144901, New Brunswick, New Jersey
  - COLUMBIA University Medical Center /ID# 149037, New York, New York
  - Cleveland Clinic Main Campus /ID# 144885, Cleveland, Ohio
  - Oregon Health and Science University /ID# 149774, Portland, Oregon
  - Vanderbilt Univ Med Ctr /ID# 144898, Nashville, Tennessee
  - Kerwin Research Center /ID# 144904, Dallas, Texas
  - McGovern Medical School /ID# 149236, Houston, Texas
  - Central Texas Neurology Consul /ID# 167417, Round Rock, Texas
- Australia (5):
  - Westmead Hospital /ID# 154403, Westmead, New South Wales
  - Q-Pharm Pty Limited /ID# 154410, Herston, Queensland
  - Royal Adelaide Hospital /ID# 153157, Adelaide, South Australia
  - Alfred Hospital /ID# 153158, Melbourne, Victoria
  - Neurodegenerative Disorders Re /ID# 153770, West Perth, Western Australia
- Canada (5):
  - University of Calgary /ID# 154393, Calgary, Alberta
  - OCT Research ULC /ID# 169688, Kelowna, British Columbia
  - Toronto Western Hospital /ID# 152818, Toronto, Ontario
  - Crchum /Id# 152819, Montreal, Quebec
  - Montreal Neurological Institut /ID# 156413, Montreal, Quebec
- France (6):
  - Hopital Universitaire Purpan /ID# 153152, Toulouse, Haute-Garonne
  - Hopital de la Timone /ID# 153113, Marseille, Provence-Alpes-Côte d'Azur Region
  - Chu de Bordeaux Hopital /Id# 153151, Bordeaux
  - Hopital B Roger Salengro /ID# 153943, Lille
  - Hopital Pitie Salpetriere /ID# 153942, Paris
  - CHU Strasbourg Hautepierre Hos /ID# 206942, Strasbourg
- Germany (5):
  - St. Josef-Hospital /ID# 201984, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 201761, Leipzig, Saxony
  - Universitaetsklinikum Ulm /ID# 153155, Ulm, Thuringia
  - KH Agatharied /ID# 154166, Hausham
  - TU Uniklinik Munchen /ID# 153154, Munich
- Italy (7):
  - Universita di Catanzaro Magna Graecia /ID# 166322, Catanzaro, Calabria
  - Policlinico Agostino Gemelli /ID# 153104, Rome, Lazio
  - IBD Center - IRCCS Istituto Clinico Humanitas /ID# 155092, Rozzano, Milano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 201982, Milan
  - Istituto Neuro Mediterraneo IR /ID# 153106, Pozzilli
  - A.O. Santa Maria /ID# 153102, Terni
  - IRCCS Ospedale San Camillo /ID# 153101, Venezia LIDO
- Japan (9):
  - National Hospital Organization Higashinagoya National Hospital /ID# 201514, Nagoya, Aichi-ken
  - National Hospital Organization Asahikawa Medical Center /ID# 201585, Asahikawa, Hokkaido
  - National Hospital Organization Utano National Hospital /ID# 201979, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 202307, Sendai, Miyagi
  - NHO Sendai Nishitaga National Hospital /ID# 202132, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital /ID# 201680, Niigata, Niigata
  - Osaka University Hospital /ID# 201980, Suita-shi, Osaka
  - Juntendo University Hospital /ID# 200870, Bunkyo-ku, Tokyo
  - National Center of Neurology and Psychiatry /ID# 202037, Kodaira, Tokyo
- Spain (2):
  - Hospital General Universitario Gregorio Maranon /ID# 200876, Madrid
  - Hosp Univ Virgen del Rocio /ID# 201039, Seville

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Hoglinger GU, Litvan I, Mendonca N, Wang D, Zheng H, Rendenbach-Mueller B, Lon HK, Jin Z, Fisseha N, Budur K, Gold M, Ryman D, Florian H; Arise Investigators. Safety and efficacy of tilavonemab in progressive supranuclear palsy: a phase 2, randomised, placebo-controlled trial. Lancet Neurol. 2021 Mar;20(3):182-192. doi: 10.1016/S1474-4422(20)30489-0. PMID 33609476

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants; one participant in the ABBV-8E12 2000 mg dose group never received study drug
Groups:
- ABBV-8E12 2000mg; ABBV-8E12 4000mg: Intravenous infusions at Day 1, Day 15, and Day 29, then every 28 days for 52 weeks; 300 mg/15 mL (participants in countries other than Japan or Spain); 1000 mg/10 mL (for participants in Japan or Spain)
Period: Overall Study
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Started | 126 | 127 | 125
Completed | 50 | 52 | 48
Not Completed | 76 | 75 | 77
Not completed — Adverse Event | 7 | 9 | 7
Not completed — Withdrew consent | 6 | 8 | 10
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Other, not specified | 62 | 58 | 58

BASELINE CHARACTERISTICS:
Population: Safety dataset: all randomized participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg | Total
Number analyzed (Participants) | 126 | 126 | 125 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (6.22) | 68.3 (7.25) | 70.0 (6.85) | 68.8 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 56 | 158
  Male | 73 | 77 | 69 | 219
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 109 | 106 | 109 | 324
  Black or African American | 0 | 1 | 1 | 2
  Asian | 17 | 17 | 15 | 49
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Multiple | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 52 in Progressive Supranuclear Palsy Rating Scale (PSPRS) Total Score
Description: The PSPRS consists of 28 items grouped in six domains: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. Items are scored on a 0 to 4 scale, except for six items that are scored on a 0 to 2 scale, with the total score ranging from 0 to 100. Higher scores indicate more severe disability or movement abnormality. Positive changes in score indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: ITT dataset: all randomized participants who received at least one dose of study drug and those with available data at baseline and at Week 52
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 59 | 56 | 59
units on a scale | 10.5 (0.94) | 10.5 (0.96) | 11.4 (0.94)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — The primary efficacy analysis utilized a likelihood-based, mixed-effects model, repeated measures (MMRM) analysis of the change from baseline for each postbaseline value and compared each ABBV-8E12 dose group with the placebo group. The model, which used all observed data, included fixed, categorical effects for treatment, site, visit, baseline score-by-visit interaction and treatment-by-visit interaction, with continuous fixed covariates for the corresponding baseline score; p = 0.998, Mixed-effects model, repeated measures; LS Mean Difference = 0.0, 95% CI 2-sided [-2.63 to 2.63], Standard Error of Mean 1.34 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.464, Mixed-effects model, repeated measures; LS Mean Difference = 1.0, 95% CI 2-sided [-1.63 to 3.58], Standard Error of Mean 1.32 — ABBV-8E12 4000 mg - Placebo

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs) are defined as any event that began or worsened in severity from first dose of study drug until 20 weeks after the last dose. For more details on AEs please see the Adverse Event section.
Time Frame: From the first dose of study drug until 20 weeks following discontinuation of study drug administration have elapsed (approximately 5 half-lives), up to 80 weeks
Population: Safety Dataset: all randomized participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 126 | 126 | 125
Participants | 108 | 111 | 111

3. Secondary Outcome: Mean Change From Baseline to Week 52 in Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions related to Activities of Daily Living, and ranges from 0-52. Higher scores are associated with more disability. Positive changes in score indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 63 | 60 | 60
units on a scale | 5.6 (0.62) | 5.8 (0.63) | 7.0 (0.63)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — The analysis utilized a likelihood-based, mixed-effects model, repeated measures (MMRM) analysis of the change from baseline for each postbaseline value and compared each ABBV-8E12 dose group with the placebo group. The model, which used all observed data, included fixed, categorical effects for treatment, site, visit, baseline score-by-visit interaction and treatment-by-visit interaction, with continuous fixed covariates for the corresponding baseline score; p = 0.812, Mixed-effects model, repeated measures; LS Mean Difference = 0.2, 95% CI 2-sided [-1.52 to 1.93], Standard Error of Mean 0.88 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.104, Mixed-effects model, repeated measures; LS Mean Difference = 1.4, 95% CI 2-sided [-0.30 to 3.16], Standard Error of Mean 0.88 — ABBV-8E12 4000 mg - Placebo

4. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Score at Week 52
Description: The Clinical Global Impression of Change (CGI-C) score is a clinician's rating scale for assessing Global Improvement of Change. The CGI-C rates improvement by 7 categories: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), very much worse (7). The CGI-C score ranges from 1 to 7, with lower scores indicating improvement.
Time Frame: Week 52
Population: ITT dataset: all randomized participants who received at least one dose of study drug and those with available data at Week 52
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 50 | 48 | 51
units on a scale | 5.1 (0.11) | 5.1 (0.11) | 5.0 (0.11)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.756, Mixed-effects model, repeated measures; LS Mean Difference = -0.0, 95% CI 2-sided [-0.36 to 0.26], Standard Error of Mean 0.16 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.409, Mixed-effects model, repeated measures; LS Mean Difference = -0.1, 95% CI 2-sided [-0.44 to 0.18], Standard Error of Mean 0.16 — ABBV-8E12 4000 mg - Placebo

5. Secondary Outcome: Mean Change From Baseline to Week 52 in Midbrain Atrophy As Measured by Volumetric Magnetic Resonance Imaging (MRI)
Description: Magnetic resonance imaging (MRI) of several different brain regions was performed and volumetric analysis was conducted to quantify midbrain atrophy. Negative changes in values indicate a reduction in volume.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 53 | 55 | 54
mm^3 | -122.0 (9.64) | -129.1 (9.69) | -128.3 (9.69)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.597, Mixed-effects model, repeated measures; LS Mean Difference = -7.2, 95% CI 2-sided [-33.86 to 19.53], Standard Error of Mean 13.54 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.642, Mixed-effects model, repeated measures; LS Mean Difference = -6.3, 95% CI 2-sided [-33.04 to 20.42], Standard Error of Mean 13.56 — ABBV-8E12 4000 mg - Placebo

6. Secondary Outcome: Mean Change From Baseline to Week 52 in Schwab and England Activities of Daily Living Scale (SEADL)
Description: The Schwab and England Activities of Daily Living (SEADL) consists of ten items intended to evaluate the daily life activities of a participant. The SEADL is composed of two sections: the first is a self-reported questionnaire in which participants grade their own daily life activities, such as dressing, using the toilet, resting, eating, and social activities (subjective assessment), and the second is an assessment of motor functions, such as postural balance, speaking, rigidity, and tremors, conducted by a clinician (objective assessment). It is a percentage scale divided into deciles, and the results are reported between 0% (bedridden) and 100% (healthy). Negative changes in values indicate a decline in health.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of independence
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 58 | 56 | 60
percentage of independence | -20.6 (1.79) | -18.0 (1.82) | -20.5 (1.77)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.323, Mixed-effects model, repeated measures; LS Mean Difference = 2.5, 95% CI 2-sided [-2.48 to 7.51], Standard Error of Mean 2.53 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.974, Mixed-effects model, repeated measures; LS Mean Difference = 0.1, 95% CI 2-sided [-4.86 to 5.02], Standard Error of Mean 2.51 — ABBV-8E12 4000 mg - Placebo

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for ABBV-8E12
Description: The maximum observed serum concentration after the first and the fifth doses in Cohort 1 and Cohort J1 was determined.
Time Frame: First Dosing Interval, 2 weeks, Day 1-14; Fifth Dosing Interval, 4 weeks, Day 85-113
Population: Participants in Cohort 1 and Cohort J1 with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Cohort 1, ABBV-8E12 2000 mg: First 30 participants enrolled into the global study from countries other than Japan who received augmented safety and PK assessments and ABBV-8E12 at a dose of 2000 mg
- Cohort 1, ABBV-8E12 4000 mg: First 30 participants enrolled into the global study from countries other than Japan who received augmented safety and PK assessments and ABBV-8E12 at a dose of 4000 mg
- Cohort J1, ABBV-8E12 2000 mg: First 9 participants enrolled into the study from Japan who received augmented safety and PK assessments and ABBV-8E12 at a dose of 2000 mg
- Cohort J1, ABBV-8E12 4000 mg: First 9 participants enrolled into the study from Japan who received augmented safety and PK assessments and ABBV-8E12 at a dose of 4000 mg
Arm/Group | Cohort 1, ABBV-8E12 2000 mg | Cohort 1, ABBV-8E12 4000 mg | Cohort J1, ABBV-8E12 2000 mg | Cohort J1, ABBV-8E12 4000 mg
Number analyzed (Participants) | 11 | 9 | 3 | 3
µg/mL
  First Dosing Interval, 2 weeks, Day 1-14 | 714 (32) | 1450 (20) | 853 (6) | 1580 (13)
  Fifth Dosing Interval, 4 weeks, Day 85-113: number analyzed (Participants) | 9 | 7 | 2 | 2
  Fifth Dosing Interval, 4 weeks, Day 85-113 | 1070 (56) | 2350 (23) | 1010 (21) | 1960 (15)

8. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) for ABBV-8E12
Description: The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax, the maximum plasma concentration. Tmax was measured after the first and the fifth doses in Cohort 1 and Cohort J1.
Time Frame: First Dosing Interval, 2 weeks, Day 1-14; Fifth Dosing Interval, 4 weeks, Day 85-113
Population: Participants in Cohort 1 and Cohort J1 with available data
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, ABBV-8E12 2000 mg | Cohort 1, ABBV-8E12 4000 mg | Cohort J1, ABBV-8E12 2000 mg | Cohort J1, ABBV-8E12 4000 mg
Number analyzed (Participants) | 11 | 9 | 3 | 3
hours
  First Dosing Interval, 2 weeks, Day 1-14 | 4.0 [3.2 to 6.1] | 4.1 [3.2 to 5.6] | 5.0 [4.0 to 5.2] | 4.8 [4.3 to 4.9]
  Fifth Dosing Interval, 4 weeks, Day 85-113: number analyzed (Participants) | 9 | 7 | 2 | 2
  Fifth Dosing Interval, 4 weeks, Day 85-113 | 3.6 [2.9 to 5.5] | 4.0 [3.3 to 46.2] | 5.0 [4.4 to 5.7] | 3.4 [3.2 to 3.5]

9. Secondary Outcome: Area Under the Concentration Time Curve (AUC) for ABBV-8E12
Description: The area under the plasma concentration-time curve (AUC; measured in µg•day/mL) is a method of measurement to determine the total exposure of a drug in blood plasma. The AUC24 of ABBV-8E12 was estimated using non-compartmental methods after the first and the fifth doses in Cohort 1 and Cohort J1.
Time Frame: First Dosing Interval, 2 weeks, Day 1-14; Fifth Dosing Interval, 4 weeks, Day 85-113
Population: Participants in Cohort 1 and Cohort J1 with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•day/mL
Arm/Group | Cohort 1, ABBV-8E12 2000 mg | Cohort 1, ABBV-8E12 4000 mg | Cohort J1, ABBV-8E12 2000 mg | Cohort J1, ABBV-8E12 4000 mg
Number analyzed (Participants) | 11 | 9 | 3 | 3
µg•day/mL
  First Dosing Interval, 2 weeks, Day 1-14 | 5070 (25) | 10400 (21) | 5950 (12) | 10400 (11)
  Fifth Dosing Interval, 4 weeks, Day 85-113: number analyzed (Participants) | 10 | 8 | 3 | 3
  Fifth Dosing Interval, 4 weeks, Day 85-113 | 13900 (28) | 31600 (36) | 15200 (21) | 23900 (15)

10. Secondary Outcome: Serum Concentration of ABBV-8E12 Prior to Infusion of a Day of Dosing (Ctrough)
Description: The concentration of ABBV-8E12 immediately prior to infusion of the fifth dose (Ctrough; measured in µg/mL) was estimated using non-compartmental methods in Cohort 1 and Cohort J1.
Time Frame: First day of the Fifth Dosing Interval, Day 85
Population: Participants in Cohort 1 and Cohort J1 with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1, ABBV-8E12 2000 mg | Cohort 1, ABBV-8E12 4000 mg | Cohort J1, ABBV-8E12 2000 mg | Cohort J1, ABBV-8E12 4000 mg
Number analyzed (Participants) | 10 | 8 | 3 | 3
µg/mL | 353 (27) | 657 (45) | 345 (32) | 595 (16)

11. Secondary Outcome: Mean Change From Baseline to Week 52 in Clinical Global Impression of Severity (CGI-S) Score
Description: The CGI-S is a clinician's rating of disease severity. The CGI-S rates severity of illness on a 7-point scale, using a range of responses from 1 (normal) through 7 (the most severely ill). This rating is based upon observed and reported symptoms, behavior, and function in the past 7 days. Positive changes in score indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 50 | 48 | 51
units on a scale | 0.6 (0.10) | 0.6 (0.10) | 0.6 (0.10)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.761, Mixed-effects model, repeated measures; LS Mean Difference = -0.0, 95% CI 2-sided [-0.31 to 0.23], Standard Error of Mean 0.14 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.678, Mixed-effects model, repeated measures; LS Mean Difference = -0.1, 95% CI 2-sided [-0.32 to 0.21], Standard Error of Mean 0.13 — ABBV-8E12 4000 mg - Placebo

12. Secondary Outcome: Mean Change From Baseline to Week 52 in Progressive Supranuclear Palsy Health Related Quality of Life Scale (PSP-QoL) Total Score
Description: The PSP-QoL is a validated patient-reported outcome measure, specifically designed to assess the quality of life of participants with PSP. There are 45 items and two subscales: physical and mental impact. Items are scored from 0 (no problem) to 4 (extreme problems). The total subscale sum scores are linearly converted into a 0 to 100 scale, and higher scores indicate a lower quality of life. Positive changes in score indicate a decline in quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 62 | 59 | 60
units on a scale | 9.2 (1.63) | 10.3 (1.65) | 10.0 (1.64)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.653, Mixed-effects model, repeated measures; LS Mean Difference = 1.0, 95% CI 2-sided [-3.50 to 5.57], Standard Error of Mean 2.30 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.748, Mixed-effects model, repeated measures; LS Mean Difference = 1.0, 95% CI 2-sided [-3.50 to 5.57], Standard Error of Mean 2.30 — ABBV-8E12 4000 mg - Placebo

13. Secondary Outcome: Mean Change From Baseline to Week 52 in Progressive Supranuclear Palsy Staging System Score (PSP-SS) Score
Description: The Progressive Supranuclear Palsy Rating Scale (PSPRS) consists of 28 items grouped in six domains: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. Items are scored on a 0 to 4 scale, except for four items that are scored on a 0 to 2 scale, with the total score ranging from 0 to 100. Higher scores indicate more severe disability or movement abnormality. The PSP-SS score is a composite of the dysphagia and gait items from the PSPRS. Positive changes in score indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 59 | 57 | 59
units on a scale | 0.8 (0.24) | 0.9 (0.24) | 1.0 (0.24)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.828, Mixed-effects model, repeated measures; LS Mean Difference = 0.1, 95% CI 2-sided [-0.60 to 0.74], Standard Error of Mean 0.34 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.543, Mixed-effects model, repeated measures; LS Mean Difference = 0.2, 95% CI 2-sided [-0.46 to 0.87], Standard Error of Mean 0.34 — ABBV-8E12 4000 mg - Placebo

14. Secondary Outcome: Mean Change From Baseline to Week 52 in Third Ventricle Atrophy As Measured by Volumetric Magnetic Resonance Imaging (MRI)
Description: Magnetic resonance imaging (MRI) of several different brain regions was performed and volumetric analysis was conducted to quantify third ventricle atrophy. Positive changes in values indicate an increase in volume.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 54 | 58 | 53
mm^3 | 157.9 (18.27) | 152.4 (18.04) | 125.0 (18.57)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.829, Mixed-effects model, repeated measures; LS Mean Difference = -5.5, 95% CI 2-sided [-55.66 to 44.63], Standard Error of Mean 25.44 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.206, Mixed-effects model, repeated measures; LS Mean Difference = -32.9, 95% CI 2-sided [-83.94 to 18.23], Standard Error of Mean 25.92 — ABBV-8E12 4000 mg - Placebo

15. Secondary Outcome: Mean Change From Baseline to Week 52 in Superior Cerebellar Peduncle Atrophy As Measured by Volumetric Magnetic Resonance Imaging (MRI)
Description: Magnetic resonance imaging (MRI) of several different brain regions was performed and volumetric analysis was conducted to quantify Superior cerebellar peduncle atrophy. Negative changes in values indicate a reduction in volume.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 51 | 55 | 54
mm^3 | -8.3 (2.78) | -4.3 (2.74) | -3.7 (2.74)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.304, Mixed-effects model, repeated measures; LS Mean Difference = 4.0, 95% CI 2-sided [-3.65 to 11.65], Standard Error of Mean 3.88 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.243, Mixed-effects model, repeated measures; LS Mean Difference = 4.5, 95% CI 2-sided [-3.11 to 12.19], Standard Error of Mean 3.88 — ABBV-8E12 4000 mg - Placebo

16. Secondary Outcome: Mean Change From Baseline to Week 52 in Brainstem Atrophy As Measured by Volumetric Magnetic Resonance Imaging (MRI)
Description: Magnetic resonance imaging (MRI) of several different brain regions was performed and volumetric analysis was conducted to quantify brainstem atrophy. Negative changes in values indicate a reduction in volume.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 48 | 49 | 43
mm^3 | -374.5 (38.42) | -400.9 (38.60) | -341.3 (40.61)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.625, Mixed-effects model, repeated measures; LS Mean Difference = -26.4, 95% CI 2-sided [-132.76 to 79.94], Standard Error of Mean 53.86 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.550, Mixed-effects model, repeated measures; LS Mean Difference = 33.2, 95% CI 2-sided [-76.34 to 142.71], Standard Error of Mean 55.47 — ABBV-8E12 4000 mg - Placebo

17. Secondary Outcome: Mean Change From Baseline to Week 52 in Whole Brain Atrophy As Measured by Volumetric Magnetic Resonance Imaging (MRI)
Description: Magnetic resonance imaging (MRI) of several different brain regions was performed and volumetric analysis was conducted to quantify whole brain atrophy. Negative changes in values indicate a reduction in volume.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 45 | 46 | 49
mm^3 | -22496.2 (1793.36) | -20757.1 (1783.00) | -18811.3 (1740.72)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.488, Mixed-effects model, repeated measures; LS Mean Difference = 1739.1, 95% CI 2-sided [-3201.75 to 6680.02], Standard Error of Mean 2502.95 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.140, Mixed-effects model, repeated measures; LS Mean Difference = 3684.9, 95% CI 2-sided [-1225.46 to 8595.29], Standard Error of Mean 2487.32 — ABBV-8E12 4000 mg - Placebo

18. Secondary Outcome: Mean Change From Baseline to Week 52 in Frontal Lobe Atrophy As Measured by Volumetric Magnetic Resonance Imaging (MRI)
Description: Magnetic resonance imaging (MRI) of several different brain regions was performed and volumetric analysis was conducted to quantify frontal lobe atrophy. Positive changes in values indicate an increase in volume.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
Number analyzed (Participants) | 48 | 49 | 43
mm^3 | 1052.6 (425.55) | 1260.5 (423.96) | 1186.1 (445.18)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 2000mg; ABBV-8E12 2000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.726, Mixed-effects model, repeated measures; LS Mean Difference = 207.9, 95% CI 2-sided [-962.98 to 1378.88], Standard Error of Mean 592.68 — ABBV-8E12 2000 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 4000mg; ABBV-8E12 4000 mg vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.828, Mixed-effects model, repeated measures; LS Mean Difference = 133.6, 95% CI 2-sided [-1075.26 to 1342.40], Standard Error of Mean 611.91 — ABBV-8E12 4000 mg - Placebo

19. Secondary Outcome: Time to Loss of Ability to Walk Independently as Measured by Progressive Supranuclear Palsy Rating Scale (PSPRS) Item 26
Description: The PSPRS consists of 28 items grouped in six domains: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. Items are scored on a 0 to 4 scale, except for six items that are scored on a 0 to 2 scale, with the total score ranging from 0 to 100. Higher scores indicate more severe disability or movement abnormality. Item 26 pertains to gait, scored as either 0 (normal); 1 (slightly wide-based or irregular or slight pulsion on turns); 2 (must walk slowly or occasionally use walls or helper to avoid falling, especially on turns); 3 (must use assistance all or almost all the time); or 4 (unable to walk, even with walker; may be able to transfer).
Time Frame: From Baseline to Week 52
Population: ITT dataset: all randomized participants who received at least one dose of study drug with available data
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | ABBV-8E12 2000 mg | ABBV-8E12 4000 mg
Number analyzed (Participants) | 126 | 126 | 125
days | 169.0 [89.0 to 255.0] | 170.0 [87.0 to 253.0] | 203.0 [169.0 to 255.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 20 weeks following discontinuation of study drug administration have elapsed (approximately 5 half-lives), up to 80 weeks. In addition, serious adverse events and protocol-related nonserious adverse events were collected from the time the participant signed the study-specific informed consent.
Description: TEAEs and TESAEs are defined as any AE or TESAE with onset or worsening reported by a participant from the time that the first dose of study is administered until 20 weeks (approximately 5 half-lives) have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Placebo | ABBV-8E12 2000mg | ABBV-8E12 4000mg
All-Cause Mortality (participants affected / at risk) | 8/126 | 9/126 | 9/125
Serious Adverse Events (participants affected / at risk) | 33/126 | 29/126 | 34/125
Other Adverse Events (participants affected / at risk) | 83/126 | 75/126 | 80/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=126) | ABBV-8E12 2000mg (N=126) | ABBV-8E12 4000mg (N=125)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
EYE SWELLING (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
GASTROINTESTINAL HYPERMOTILITY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 2 (2) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 1 (1)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 2 (2)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 4 (4) | 1 (1) | 3 (4)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 1 (2)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 6 (7) | 5 (7) | 6 (7)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FOREIGN BODY ASPIRATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
RESIDUAL URINE VOLUME (Investigations) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
BRAIN MIDLINE SHIFT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
PROGRESSIVE SUPRANUCLEAR PALSY (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HYGROMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
BLADDER OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
MICTURITION DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=126) | ABBV-8E12 2000mg (N=126) | ABBV-8E12 4000mg (N=125)
CONSTIPATION (Gastrointestinal disorders) | 7 (7) | 9 (12) | 6 (6)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 10 (10) | 8 (10)
FATIGUE (General disorders) | 2 (9) | 9 (19) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9) | 5 (5) | 6 (9)
URINARY TRACT INFECTION (Infections and infestations) | 14 (19) | 13 (14) | 18 (28)
CONTUSION (Injury, poisoning and procedural complications) | 17 (23) | 16 (20) | 23 (30)
FALL (Injury, poisoning and procedural complications) | 43 (96) | 37 (70) | 48 (85)
SKIN ABRASION (Injury, poisoning and procedural complications) | 15 (27) | 11 (16) | 8 (9)
SKIN LACERATION (Injury, poisoning and procedural complications) | 19 (29) | 17 (19) | 21 (26)
WEIGHT DECREASED (Investigations) | 11 (12) | 10 (12) | 13 (15)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 8 (8)
DIZZINESS (Nervous system disorders) | 2 (2) | 8 (9) | 4 (4)
HEADACHE (Nervous system disorders) | 8 (13) | 9 (11) | 4 (4)
ANXIETY (Psychiatric disorders) | 7 (8) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 8 (8) | 10 (12) | 3 (3)
INSOMNIA (Psychiatric disorders) | 5 (6) | 6 (8) | 8 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 5 (6) | 5 (5)
RASH (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT02985879/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT02985879/SAP_001.pdf